CLINICAL TRIAL: NCT00236912
Title: A Multi-center, Open-label, Randomized Study to Compare the Safety and Efficacy of Once Daily Levofloxacin Along With Once Daily Metronidazole Versus Piperacillin/Tazobactam in the Treatment of Complicated Appendicitis
Brief Title: A Study Comparing Safety and Efficacy of Levofloxacin and Metronidazole Versus Piperacillin/Tazobactam in Treating Complicated Appendicitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was terminated due to low enrollment.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002656
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Appendicitis
Keywords: complicated appendicitis; antibiotics; appendicitis; infection
MeSH Terms: conditions — Appendicitis; Infections | interventions — Levofloxacin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: levofloxacin; metronidazole

SUMMARY:
The purpose of this study is to compare the efficacy and safety of two treatment regimens in treating patients with complicated appendicitis. Appendicitis requires antibiotic treatment when the appendix ruptures (complicated appendicitis). This is a study comparing intravenous (IV) antibiotic therapy of levofloxacin/metronidazole versus piperacillin/tazobactam for 4 to 14 days. Patients may be switched to oral therapy after 48 hours, at the doctor's discretion.

DETAILED DESCRIPTION:
Appendicitis may be classified as uncomplicated (the appendix has not ruptured) or complicated (the appendix has ruptured or gangrene has begun). Typically all patients with complicated appendicitis are treated with intravenous (IV, through a vein) antibiotic therapy. This is a multicenter, open-label, randomized study of patients who have complicated appendicitis. Prior to surgery, patients will be randomized to either the levofloxacin/metronidazole IV group (given once daily) or the piperacillin/tazobactam IV group (given 4 times daily) and will be started on study drug. Patients who are confirmed during surgery to have complicated appendicitis, will continue to receive study drug to complete a total of 4-14 days of therapy. Those found to have uncomplicated appendicitis will stop taking study drug and be discontinued from the study. Patients may be switched after 48 hours to oral therapy, at the doctor's discretion. Patients randomized to levofloxacin/metronidazole will be switched to oral levofloxacin/metronidazole given once daily. Patients randomized to piperacillin/tazobactam will be switched to oral amoxicillin/clavulanate acid given twice daily. While in the hospital, daily assessments will be made of the patient for clinical signs and symptoms of post-operative wound infection. In addition, temperature, vital signs, pertinent physical findings, white blood count (until normal), and tests for infection will be assessed daily while in the hospital. Wound assessments and laboratory tests will be performed on the last visit as an outpatient. The main objective of this study is to determine the safety and effectiveness of the regimen containing levofloxacin and metronidazole compared with the regimen of piperacillin/tazobactam in the treatment of complicated appendicitis.

Levofloxacin 750 mg IV (through a vein) or orally then metronidazole 1500 milligrams IV (or tablet form by mouth) once daily for 4 to 14 days; or piperacillin/tazobactam 3.375 grams IV every 6 hours (or amoxicillin/clavulanate acid 875/125 milligram tablets by mouth every 12 hours) for 4 to 14 days

ELIGIBILITY:
Inclusion Criteria:

* Two or more symptoms of acute appendicitis for at least 24 hours or radiologic evidence of complicated appendicitis
* Able to take medicine orally after recovering from surgery
* If female, using birth control

Exclusion Criteria:

* History of allergy to any study medication
* Life expectancy < 72 hours
* APACHE II (health) score > 25
* Neutropenic (low white blood cell count)
* HIV positive with current or past CD4 count < 200/mm^3
* Low platelet count (bleeds easily)
* Malnourished with low albumin
* Condition requiring use of major tranquilizers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2003-07; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Clinical success at the post-therapy visit; safety by adverse events.

SECONDARY OUTCOMES:
Clinical and microbiologic response at post-therapy and post-study; costs associated with care.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Multicenter, Open-Label, Randomized Study to Compare the Safety and Efficacy of Once Daily Levofloxacin Along With Once Daily Metronidazole Versus Piperacillin/Tazobactam in the Treatment of Complicated Appendicitis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=484&filename=CR002656_CSR.pdf